CLINICAL TRIAL: NCT03377257
Title: Efficacy and Safety of Zolmitriptan by Sublingual Administration in the Treatment of Cluster Headache: A Multi-center Randomized Cross-controlled Trial
Brief Title: Efficacy and Safety of Zolmitriptan by Sublingual Administration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Xijing-CH-zolmi
Record Dates: First submitted 2017-12-05; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-05

CONDITIONS: Cluster Headache
Keywords: Cluster headache; zolmitriptan; Sublingual administration
MeSH Terms: conditions — Cluster Headache | interventions — zolmitriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): The treatment with oral zolmitriptan is 2.5mg when headache attack.
  Interventions: Drug: zolmitriptan by oral
- Experimental group (Experimental): The treatment with zolmitriptan by sublingual administration is 2.5mg when headache attack.
  Interventions: Drug: zolmitriptan by sublingual administration

INTERVENTIONS:
Drug: zolmitriptan by sublingual administration — Experimental group
  Other Names: zolmitriptan
  Arms: Experimental group
Drug: zolmitriptan by oral — Active group
  Arms: Active group

SUMMARY:
The purpose is to evaluate the effectiveness and safety profile of zolmitriptan by Sublingual administration for the acute treatment of Cluster headache.

DETAILED DESCRIPTION:
Cluster headache is a primary neurological disorder characterized by intensive attacks and severe sharp headache, can cause a range of symptoms such as conjunctival congestion, runny nose, miosis, forehead sweat. The disability resulting from cluster headache can be severe imposing a considerable health burden upon the sufferer and society. The purpose of this study, using oral zolmitriptan as the control, is to evaluate the effectiveness and safety of zolmitriptan by sublingual administration for the acute treatment of cluster headache. Patients are asked to maintain a headache diary throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than or equal to 18 years and less than 70 years;
* The diagnosis of cluster headache is made according to The International Classification of Headache Disorders: 3rd edition (beta version)(ICHD-III β);
* Consent form signed by the participant or his/her authorized surrogate.

Exclusion Criteria:

* Patients had primary or secondary headache disorders other than cluster headache;
* Female subjects of childbearing age will be excluded if they were pregnant, lactating or planning a pregnancy in the next year or if they were not using an adequate form of birth control;
* Patients will be excluded if they had significant medical or psychiatric disease;
* Patients will be excluded if they had coronary heart disease or not suitable for the treatment of zolmitriptan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
The points-reducing of visual analogue scale several minutes after sublingual zolmitriptan tablet | 5, 10, 15 minutes after administration
  The difference of the percentage of the headache attacks whose visual analogue scale points reduce from 7-10 to 0-3 5, 10, 15 minutes after administration between sublingual and oral zolmitriptan tablet

SECONDARY OUTCOMES:
The percentage of side effects; | 3 hours
  The difference of the percentage of side effects in 3 hours after the administration between sublingual and oral zolmitriptan tablet
The percentage of discontinued the drug | 3 days
  The percentage of discontinued the drug because of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: Undecided
cluster headache